CLINICAL TRIAL: NCT00660049
Title: Feasibility Study of a Novel Device for Chronic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, Anne Chang, Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-02252008-1026; IRB Protocol #: 11074 (Other: Stanford University)
Record Dates: First submitted 2008-04-04; First posted 2008-04-17 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Ulcer; Wounds and Injuries
MeSH Terms: conditions — Ulcer; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SNaP application (Experimental): This is an "open label" pilot study of SNaP Advanced Wound Care System
  Interventions: Device: SNaP Advanced Wound Care System; Other: SNaP

INTERVENTIONS:
Device: SNaP Advanced Wound Care System — Application of negative pressure device daily per instructions
  Other Names: SNaP device (SmartNegative Pressure device)
Other: SNaP — Daily use
  Other Names: SNaP device
Other: SNaP — Daily application per protocol

SUMMARY:
The purpose of this study is to evaluate the feasibility and usability of a new portable and compact wound dressing device for the treatment of small chronic skin wounds.

DETAILED DESCRIPTION:
This is an open label study

ELIGIBILITY:
Inclusion Criteria:- Venous stasis ulcer or other chronic wound on the lower extremity that is >1.5cm and <10cm at widest point

* The wound must have at least 2 cm of intact epithelium surrounding it.
* A wound such as a pressure ulcer or chronic ulcer on a location other than the lower extremity may also be included in the study if it meets the size requirements and a reliable seal can be achieved.
* Ulcer must not have healed for >14 days under standard treatment.
* Chronic wound with prior graft placement will be allowed in the study.
* Patient is >18 years old.
* Willing and able to sign informed consent.

Exclusion Criteria:- Active wound infection.

* 3+ or greater pitting edema of lower extremity
* History of malignancy at wound site. However, wounds that are closing by secondary intent after surgical clearance of prior tumor will be allowed in the study.
* Thick eschar at wound base after debridement.
* Wound location is not amenable to forming an airtight seal and placement of device.
* Ulcers due to inflammatory conditions such as pyoderma gangrenosum, rheumatoid arthritis, vasculitis, cryoglobulinemia, necrobiosis lipoidica diabeticorum, lupus or pancreatic panniculitis, cryofibrinogenemia, calcinosis cutis, scleroderma, Raynaud's syndrome.
* Current smoker (must have quit for >3 weeks)
* Wound with exposed bone, blood vessels, tendon
* Significant immunosuppression (as determined by the investigator and sponsor) such as high dose prednisone
* Fasting blood sugar >200 by study personnel administered bedside fingerstick blood glucose
* Ankle brachial index less than lower limit of normal (<0.60) as performed and determined by licensed physician (necessary only for patients with lower extremity wounds).
* Pregnancy
* Incapable of giving informed consent
* Inability to comply with study procedures including lack of telephone access for week 8 telephone survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-03; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Anne Lynn S. Chang, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No sharing

REFERENCES:
- [Background] Fong KD, Hu D, Eichstadt SL, Gorell E, Munoz CA, Lorenz HP, Chang AL. Initial clinical experience using a novel ultraportable negative pressure wound therapy device. Wounds. 2010 Sep;22(9):230-6. PMID 25901554

RESULTS

PARTICIPANT FLOW:
Groups:
- SNaP Application: This is an "open label" pilot study of SMart Negative Pressure (SNaP) Advanced Wound Care System
  SNaP Advanced Wound Care System: Application of negative pressure device daily per instructions
  SNaP: Daily use
  SNaP: Daily application per protocol
Period: Overall Study
Arm/Group | SNaP Application
Started | 12
Completed | 6
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: 12
Groups:
- Open Label Single Arm Study: Eligible participants
Arm/Group | Open Label Single Arm Study
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 55 [18 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Ease of Use for Patients
Description: Participants were given instructions to use the SNaP device home. Participants completed a questionnaire reporting whether the device was easy to use, worthwhile to use, and whether they would use the device again. Numbers responding positively to each question are presented.
Time Frame: Baseline up to 31 days
Population: All participants
Measure: Number; unit: participants
Groups:
- Open Label Single Arm Study: All participants who use the device
Arm/Group | Open Label Single Arm Study
Number analyzed (Participants) | 12
participants
  Easy to use | 8
  Worthwhile to use | 10
  I would use this device again | 9

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Eligible Participants: This is an "open label" pilot study of SNaP Advanced Wound Care System
  SNaP Advanced Wound Care System: Application of negative pressure device daily per instructions
  SNaP: Daily use
  SNaP: Daily application per protocol
Arm/Group | Eligible Participants
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Eligible Participants (N=12)
wound pain (Skin and subcutaneous tissue disorders) | 3
ipsilateral knee pain (Musculoskeletal and connective tissue disorders) | 3/11 — 11 patients that used device lower extremity were at risk

LIMITATIONS AND CAVEATS:
Open label design without comparator arm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less